CLINICAL TRIAL: NCT01943552
Title: Peri-operative Intervention With Nebulized Ipratropium Bromide in Chinese Patients With Chronic Obstructive Pulmonary Disease (COPD): a Randomized, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Trial.
Brief Title: Ipratropium Bromide in Peri-Operative COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244.2514
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2016-09-12 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

ARMS (2):
- ipratropium (Experimental): 500 mcg four times a day
  Interventions: Drug: ipratropium bromide
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — normal saline
  Arms: placebo
Drug: ipratropium bromide — ipratropium bromide
  Arms: ipratropium

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-centre trial.The trial aims to evaluate efficacy of nebulized ipratropium bromide in Chinese peri-operative patients with COPD under general anaesthesia.

ELIGIBILITY:
Inclusion criteria:

* All patients must sign an informed consent.
* Male or female patients aged >= 40 years and <= 80 years
* All patients must be diagnosed with COPD and must meet the following spirometric criterion: post-bronchodilator forced expiratory volume in 1 second (FEV1) < 70% of forced vital capacity (FVC) at Screening Visit (Visit 1).
* All patients have relatively stable COPD (i.e. have no COPD exacerbation within 4 weeks prior to Screening Visit).
* All patients are about to receive selective surgical procedures of lobectomy or right bilobectomy or segmentectomy under general anaesthesia, whilst the estimated time of surgical procedures lasts for not less than 2 hours, and the estimated time of general anaesthesia lasts for not less than 3 hours and not longer than 5 hours.
* Patients must be able to perform all study related procedures including technically acceptable pulmonary function tests (PFTs).

Exclusion criteria:

* Patients who need maintenance treatment of bronchodilators (including anticholinergics, ß-agonists, xanthines).
* Patients with a recent history (i.e. six months or less) of myocardial infarction
* Patients with any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year
* Patients with symptomatic chronic heart failure (i.e. New York Heart Association functional class III-IV)
* Known narrow angle glaucoma
* Patients with prostatic hyperplasia or bladder neck obstruction with significant symptoms
* Patients with a history of asthma, allergic rhinitis or who have a blood eosinophil count >= 600 / mm3 (0.6×10^9/L). A repeat eosinophil count will not be conducted in these patients

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- China (9):
  - 244.2514.86008 Boehringer Ingelheim Investigational Site, Chengdu
  - 244.2514.86006 Boehringer Ingelheim Investigational Site, Guangzhou
  - 244.2514.86007 Boehringer Ingelheim Investigational Site, Guangzhou
  - 244.2514.86010 Boehringer Ingelheim Investigational Site, Guangzhou
  - 244.2514.86009 Boehringer Ingelheim Investigational Site, Hangzhou
  - 244.2514.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 244.2514.86002 Boehringer Ingelheim Investigational Site, Tianjin
  - 244.2514.86011 Boehringer Ingelheim Investigational Site, Wuhan
  - 244.2514.86012 Boehringer Ingelheim Investigational Site, Wuhan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 192 patients were randomized in a 1:1 ratio(96 patients in each group).1 patient each in both treatment groups did not receive the treatment.1 patient, who was randomized to the placebo group, but received nebulized ipratropium bromide, so the actual numbers of patients received nebulized ipratropium bromide and placebo were 96 and 94 respectively
Pre-assignment Details: This was randomised, double-blind, placebo-controlled, parallel-group, multicentre trial which aims to evaluate efficacy and safety of nebulized ipratropium bromide in Chinese peri-operative patients with chronic obstructive pulmonary disease (COPD) under general anaesthesia.
Groups:
- Nebulized Ipratropium Bromide: 500 microgram (mcg) ipratropium bromide solution was administered orally via nebulizer four times a day up to 11 days.
- Placebo: 4 milliliter (ml) normal saline was administered orally via nebulizer four times a day up to 11 days.
Period: Overall Study
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Started | 96 (One patient was randomised to the placebo group, but received nebulized ipratropium bromide.) | 94
Completed | 71 | 69
Not Completed | 25 | 25
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Other Reasons | 16 | 17

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized Ipratropium Bromide | Placebo | Total
Number analyzed (Participants) | 96 | 94 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (6.5) | 62.4 (6.4) | 62.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 83 | 85 | 168

OUTCOME MEASURES:

1. Primary Outcome: Change of Forced Expiratory Volume in 1 Second (FEV1) From Pre-bronchodilator at Baseline to Post-nebulization One Day Before the Surgery
Description: Change of forced expiratory volume in 1 second (FEV1) from pre-bronchodilator at baseline to post-nebulization one day before the surgery (Treatment day 3). Measurements of FEV1 were performed using calibrated electronic spirometers. Equipment and techniques should conform to American Thoracic Society (ATS) criteria (P05-12782). At screening visit, pulmonary function testing (PFT) was performed at baseline and repeated 30 minutes following inhalation of 4 puffs of salbutamol hydrofluoroalkanes metered-dose inhaler (HFA MDI). At treatment day 3, pulmonary function testing was performed 60 minutes following the inhalation of investigational drug. Spirometry was conducted with the patient in a seated position having abstained from medications. The best of three efforts was defined as the highest FEV1 each obtained on any of three efforts meeting the ATS criteria and it was selected regardless of whether they came from different spirometric manoeuvres or the same manoeuvre.
Time Frame: Baseline and Treatment day 3
Population: Full analysis set (FAS): All patients in the treated set who had observed analysable data in at least one efficacy endpoint. (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 94 | 89
ml | 169.9 (29.07) | 15.0 (29.35)
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; The analysis of covariance (ANCOVA) method was used to compare the change of FEV1 from pre-bronchodilator at baseline to post-nebulization on treatment day 3 between the active arm and the placebo arm, with baseline value as covariate and two stratification factors based on acute bronchodilator responsiveness at baseline and age as main effects; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 154.9, 95% CI 2-sided [91.08 to 218.63], Standard Error of Mean 32.32 — The Mean Difference; nebulized ipratropium minus placebo was estimated by the difference of their adjusted means

2. Secondary Outcome: Change of Forced Vital Capacity (FVC) From Pre-bronchodilator at Baseline to Post-nebulization One Day Before the Surgery
Description: Change of forced vital capacity (FVC) from pre-bronchodilator at baseline to post-nebulization one day before the surgery (Treatment day 3). Measurements of FVC were performed using calibrated electronic spirometers. Equipment and techniques should conform to American Thoracic Society (ATS) criteria (P05-12782). At Visit 1, pulmonary function testing (PFT) was performed at baseline and repeated 30 minutes following inhalation of 4 puffs of salbutamol hydrofluoroalkanes metered-dose inhaler (HFA MDI). At Visit 3, pulmonary function testing was performed 60 minutes following the inhalation of investigational drug. Spirometry was conducted with the patient in a seated position having abstained from medications. The best of three efforts was defined as the highest FVC each obtained on any of three efforts meeting the ATS criteria and it was selected regardless of whether they came from different spirometric manoeuvres or the same manoeuvre.
Time Frame: Baseline and Treatment day 3
Population: Full analysis set (FAS). (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 94 | 89
ml | 59.4 (48.76) | 8.5 (49.27)
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; The analysis of covariance (ANCOVA) method was used to compare the change of forced vital capacity (FVC) from pre-bronchodilator at baseline to post-nebulization on treatment day 3 between the active arm and the placebo arm, with baseline value as covariate and two stratification factors based on acute bronchodilator responsiveness at baseline and age as main effects; Test type: Superiority or Other; p = 0.3509, ANCOVA; Mean Difference (Net) = 51.0, 95% CI 2-sided [-56.55 to 158.46], Standard Error of Mean 54.48 — The Mean Difference; nebulized ipratropium minus placebo was estimated by the difference of their adjusted means

3. Secondary Outcome: Change of Blood Gas Analyses From Pre-bronchodilator at Baseline to Post-nebulization One Day Before the Surgery: Arterial Oxygen Pressure (PaO2) Value
Description: Change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization one day before the surgery (Treatment day 3): arterial oxygen pressure (PaO2) value
Time Frame: Baseline and Treatment day 3
Population: Full analysis set (FAS). (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 89 | 80
mmHg | 3.2 (1.92) | 0.5 (1.92)
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; The analysis of covariance (ANCOVA) method was used to compare the change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization on treatment day 3 for PaO2 between the active arm and the placebo arm, with baseline value as covariate and two stratification factors based on acute bronchodilator responsiveness at baseline and age as main effects; Test type: Superiority or Other; p = 0.2069, ANCOVA; Mean Difference (Net) = 2.8, 95% CI 2-sided [-1.54 to 7.07], Standard Error of Mean 2.18 — The Mean Difference; nebulized ipratropium minus placebo was estimated by the difference of their adjusted means

4. Secondary Outcome: Change of Blood Gas Analyses From Pre-bronchodilator at Baseline to Post-nebulization One Day Before the Surgery: Oxygen Saturation
Description: Change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization one day before the surgery (Treatment day 3): Oxygen saturation
Time Frame: Baseline and Treatment day 3
Population: Full analysis set (FAS). (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: Percentage of Oxygen
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 89 | 81
Percentage of Oxygen | 0.6 (0.25) | 0.3 (0.25)
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; The analysis of covariance (ANCOVA) method was used to compare the change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization on treatment day 3 for Oxygen saturation between the active arm and the placebo arm, with baseline value as covariate and two stratification factors based on acute bronchodilator responsiveness at baseline and age as main effects; Test type: Superiority or Other; p = 0.1899, ANCOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.19 to 0.93], Standard Error of Mean 0.28 — The Mean Difference; nebulized ipratropium minus placebo was estimated by the difference of their adjusted means

5. Secondary Outcome: Change of Blood Gas Analyses From Pre-bronchodilator at Baseline to Post-nebulization One Day Before the Surgery: Arterial Carbon Dioxide Pressure (PaCO2) Value
Description: Change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization one day before the surgery (Treatment day 3): arterial carbon dioxide pressure (PaCO2) value
Time Frame: Baseline and Treatment day 3
Population: Full analysis set (FAS). (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 89 | 80
mmHg | -0.1 (0.51) | -0.5 (0.52)
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; The analysis of covariance (ANCOVA) method was used to compare the change of blood gas analyses from pre-bronchodilator at baseline to post-nebulization on treatment day 3 for PaCO2 between the active arm and the placebo arm, with baseline value as covariate and two stratification factors based on acute bronchodilator responsiveness at baseline and age as main effects; Test type: Superiority or Other; p = 0.4758, ANCOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.72 to 1.55], Standard Error of Mean 0.57 — The Mean Difference; nebulized ipratropium minus placebo was estimated by the difference of their adjusted means

6. Secondary Outcome: Main Post-operative Pulmonary Complications (Including Pneumonia, Atelectasis and Acute Respiratory Failure) Within Three Weeks After the Surgery
Description: Number of patients with at least one main post-operative pulmonary complications (including pneumonia, atelectasis and acute respiratory failure) within three weeks after the surgery. Post-operative pneumonia was defined by the presence of the following criteria: persistent lung infiltrate on chest X-ray or chest computerized tomography (CT)-scan, white blood cell count >10,000 /mm3 and fever. Post-operative atelectasis was diagnosed by presence of atelectasis affecting one lobe or several lobes in chest X-ray test or chest CT-scan. Post-operative acute respiratory failure was defined by the presence of: PaO2 < 60 mmHg and/or PaCO2 > 50 mmHg while breathing air or other evidences which were considered as respiratory failure by investigators.
Time Frame: From surgery to 3 weeks post surgery, up to 21 days
Population: Surgery complete set (SCS): All patients who completed surgery.
Measure: Number; unit: Participants
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Number analyzed (Participants) | 77 | 78
Participants | 8 | 14
Statistical Analysis 1: Comparison: Nebulized Ipratropium Bromide vs Placebo; For main post-operative pulmonary complications, the Cochran-Mantel-Haenszel analysis was performed on the SCS. Mantel-Haenszel test with strata based on acute bronchodilator responsiveness at baseline and age was used to compare the number of patients with main post-operative pulmonary complications between the two arms; Test type: Superiority or Other; p = 0.1779, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel Test Statistic = 1.82

ADVERSE EVENTS:
Time Frame: From first drug administration until 14 days after the last drug administration, up to 32 days
Arm/Group | Nebulized Ipratropium Bromide | Placebo
Serious Adverse Events (participants affected / at risk) | 5/96 | 4/94
Other Adverse Events (participants affected / at risk) | 15/96 | 16/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebulized Ipratropium Bromide (N=96) | Placebo (N=94)
Cardiac arrest (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebulized Ipratropium Bromide (N=96) | Placebo (N=94)
Post procedural pneumonia (Infections and infestations) | 2 | 9
Wound complication (Injury, poisoning and procedural complications) | 8 | 10
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Hypertension (Vascular disorders) | 5 | 1

LIMITATIONS AND CAVEATS:
192 patients were entered in this trial. It was planned to treat 96 with Ipratropium bromide and 96 with Placebo. Out of these, one patient was randomised to the placebo group, but received nebulized ipratropium bromide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.